CLINICAL TRIAL: NCT02316821
Title: RTA 402 Phase 2 Clinical Trial (A Randomized, Double-blind, Placebo-controlled Clinical Trial in Patients With Chronic Kidney Disease and Type 2 Diabetes)
Brief Title: The Phase II Study of Bardoxolone Methyl in Patients With Chronic Kidney Disease and Type 2 Diabetes; TSUBAKI Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTA 402-005
Record Dates: First submitted 2014-11-27; First posted 2014-12-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 2; Diabetic Nephropathies; Kidney Diseases; Renal Insufficiency, Chronic; Diabetes Complications; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Renal Insufficiency; Urologic Diseases; bardoxolone methyl
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Diabetes Mellitus; Diabetic Nephropathies; Kidney Diseases; Diabetes Complications; Endocrine System Diseases; Glucose Metabolism Disorders; Metabolic Diseases; Renal Insufficiency; Urologic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bardoxolone methyl (Experimental): bardoxolone methyl capsules, dosage To Be Determined, once daily for 16 weeks
  Interventions: Drug: RTA 402
- Placebo (Placebo Comparator): Placebo capsules, once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RTA 402
  Arms: bardoxolone methyl
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of RTA 402 in chronic kidney disease (CKD) patients with type 2 diabetes in a double-blind, placebo-controlled study when this compound is administered once daily for 16 weeks in an intrapatient dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

* CKD patients with type 2 diabetes mellitus
* Patients whose estimated GFR levels are eligible for this study
* Patients being treated with stable dose of angiotensin converting enzyme (ACE) inhibitors and/or angiotensin II receptor blocker (ARB) etc.

Exclusion Criteria:

* Patients with type 1 diabetes mellitus
* Patients with known non-diabetic renal disease
* Patients with a history of renal transplantation
* Patients with mean systolic blood pressure > 160 mmHg or diastolic blood pressure > 90 mmHg
* Patients with Hemoglobin A1c > 10%
* Patients with cardiovascular disease specified in the study protocol etc.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-12; Primary Completion 2016-05 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Safety: Number and types of adverse events | Up to 16 weeks
  Count of adverse events, by type, in the bardoxolone methyl arm compared to the placebo arm
Change in glomerular filtration rate (GFR) measured by inulin clearance after 16 weeks of study drug administration, compared to baseline GFR | Up to 16 weeks
  Change in GFR from baseline to 16 weeks

SECONDARY OUTCOMES:
Change in estimated GFR (eGFR) after 16 weeks of study drug administration, compared to baseline eGFR | Up to 16 weeks
  Change in eGFR from baseline to 16 weeks
Profiles of pharmacokinetics of plasma RTA 402 concentration: Trough (Pre-dose) and peak (2-4 hours post dose) concentrations of study drug at steady state | Baseline, week 2, 6, 10, and 4 weeks after completion of study treatment
  Relationship between the study drug dose and the trough (Pre-dose) and peak (2-4 hours post dose) concentrations of study drug at steady state

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Yoshioka K, Kaneko H, Haruyama W, Tomiyama T, Takami A, Kitayama T, Yamasaki K. Multi-Omics Reveal Antioxidant Effects of Bardoxolone Methyl in the Phase 2 Study of Bardoxolone Methyl in Patients with CKD and Type 2 Diabetes Study. Kidney360. 2025 Nov 1;6(11):1880-1889. doi: 10.34067/KID.0000000853. Epub 2025 Jun 11. PMID 40498549
- [Derived] Mwesigwa N, Millar Vernetti P, Kirabo A, Black B, Ding T, Martinez J, Palma JA, Biaggioni I, Kaufmann H, Shibao CA. Atomoxetine on neurogenic orthostatic hypotension: a randomized, double-blind, placebo-controlled crossover trial. Clin Auton Res. 2024 Dec;34(6):561-569. doi: 10.1007/s10286-024-01051-2. Epub 2024 Sep 19. PMID 39294522
- [Derived] Ikejiri K, Suzuki T, Muto S, Takama H, Yamawaki K, Miyazawa T, Urakawa I, Aoki Y, Otsuki A, Katsuoka F, Kinoshita K, Nangaku M, Akizawa T, Yamamoto M. Effects of NRF2 polymorphisms on safety and efficacy of bardoxolone methyl: subanalysis of TSUBAKI study. Clin Exp Nephrol. 2024 Mar;28(3):225-234. doi: 10.1007/s10157-023-02427-w. Epub 2023 Nov 14. PMID 37962746